CLINICAL TRIAL: NCT06425770
Title: Investigating the Accuracy of Conventional vs Digital Impressions and Conventional vs 3D Fabricated Casts in Capturing the Emergence Profile Around Maxillary Anterior Single Implant-supported Crowns
Brief Title: Digital vs Conventional Impression in Capturing the Emergence Profile Around Maxillary Anterior Implant-supported Crowns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 129/2023
Record Dates: First submitted 2024-05-06; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-01

CONDITIONS: Dental Implants, Single-Tooth; Dental Impression Technique
Keywords: Peri-Implant Emergence Profile; Dental Impression Technique; Dental Implants, Single-Tooth; Esthetics, Dental; Crowns; Denture, Partial, Fixed; Computer-Aided Design
MeSH Terms: interventions — POLR1G protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional cast (Active Comparator): conventional impression with elastomer (silicon), from which a high-precision epoxi-resin cast with gingival mask will be created
  Interventions: Procedure: conventional impresion and cast
- indirect digital impression and 3D printed cast (Experimental): the provisional restoration will be scanned with intraoral scanner extraorally, based on which a virtual model will be created, from which a 3D printed cast will be created with manually fabricated gingival mask based on the provisional restoration
  Interventions: Procedure: indirect digital impression and 3D printed cast
- direct digital impression (Experimental): the emergence profile will be directly scanned with intraoral scanner at 0, 2, 10, and 20 minutes after removing the provisional restoration
  Interventions: Procedure: direct digital impression

INTERVENTIONS:
Procedure: indirect digital impression and 3D printed cast — the provisional restoration will be scanned with intraoral scanner extraorally, based on which a virtual model will be created, from which a 3D printed cast will be created with manually fabricated gingival mask based on the provisional restoration
  Arms: indirect digital impression and 3D printed cast
Procedure: direct digital impression — the emergence profile will be directly scanned with intraoral scanner at 0, 2, 10, and 20 minutes after removing the provisional restoration
  Arms: direct digital impression
Procedure: conventional impresion and cast — conventional impression with elastomer (silicon), from which a high-precision epoxi-resin cast with gingival mask will be created
  Arms: conventional cast

SUMMARY:
This study compares conventional impression and cast fabrication to direct/indirect digital scannig and 3D printed casts regarding their accuracy in replicating the peri-implant emergence profile of single implants in the maxillary anterior region (FDI #15-25).

DETAILED DESCRIPTION:
Correct design of the peri-implant emergence profile (EP) is crucial for maintaining the health of the supracrestal complex and long-term success of the implant implant-prosthodontics. After its formation with a provisional restoration, its shape needs to be transferred to the final restoration via conventional elastomeric or digital (direct/indirect) impression taking.

Our aims are to investigate around maxillary anterior single implants in patients with thick gingival phenotype:

1. the accuracy of direct digital impression vs indirect digital impression vs conventional elastomeric impression in capturing the EP and implant position
2. the accuracy of 3D printed cast with conventional gingival mask vs conventional epoxy-resin cast with gingival mask in replicating the EP and implant position
3. the amount of soft tissue collapse at 0,2,10,20 minutes following the removal of the provisional restoration in case of direct EP scanning

ELIGIBILITY:
Inclusion Criteria:

* Adult above 18 yo
* No systematic deseases
* Good oral hygene (FMPS < 25%)
* Stable occlusion
* Thick phenotype
* Single missing maxilary anterior (FDI #15-25 position) tooth replaced with osseointegrated bone level impant
* Correctly formed soft tissue with CAD/CAM temporary abutment for min. 3 months
* Neighbouring teeth in place and in good condition
* Patient voluntarily accepts and signs the patient leaflets for the trial

Exclusion Criteria:

* Active periodontitis
* Peri-implant inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
3D RMS - root mean square difference | at impression taking, 0,2,10,20 mins
  The absolute mean deviation between the emergence profiles replicated with different impression techniques along the whole surface of the EP

SECONDARY OUTCOMES:
Linear vertical soft tissue change | at impression taking, 0,2,10,20 mins
  Vertical height change of the buccal gingiva marginal level measured at the mesial and distal papilae and mid-facial levels
Linear horizontal soft tissue change | at impression taking, 0,2,10,20 mins
  Horizontal thickness change of the buccal and palatal gingiva at three levels at each third of the distance between the implant platform and the marginal gingiva.
2D RMS - root mean square difference | at impression taking, 0,2,10,20 mins
  The absolute mean deviation between the emergence profiles replicated with different impression techniques along vertical and horizontal cross-sections.
Patient reported outome measures - evaluation of the impression method | at the end of each session of the digital and conventional impression taking
  Patient evaluation of the different types of impression methods on a visual analoge scale based questionnaire

OTHER OUTCOMES:
Pink esthetic score/PES | at impression taking, definitive prosthetic rehabilitation (2 weeks after impression), 6 and 12 months follow-up
  pink esthetic score of the definitive restoration
White esthetic score/WES | at impression taking, definitive prosthetic rehabilitation (2 weeks after impression), 6 and 12 months follow-up
  white esthetic score of the definitive restoration
functional implant prosthodontic score/FIPS | at impression taking, definitive prosthetic rehabilitation (2 weeks after impression), 6 and 12 months follow-up
  functional implant prosthodontic score of the definitive restoration

CONTACTS AND LOCATIONS:
Overall Officials: Krisztina Mikulás, PhD, Principal Investigator — Department of Prosthodontics, Semmelweis University
Locations (1):
- Semmelweis University, Department of Prosthodontics, Budapest, Pest County, Hungary

REFERENCES:
- [Background] Li J, Chen Z, Wang M, Wang HL, Yu H. Dynamic changes of peri-implant soft tissue after interim restoration removal during a digital intraoral scan. J Prosthet Dent. 2019 Sep;122(3):288-294. doi: 10.1016/j.prosdent.2018.07.020. Epub 2019 Mar 15. PMID 30885583
- [Background] Xiong J, Sun W, Huang B, Ji W, Shi B. Effect of the implant-supported provisional restoration on the accuracy of digital peri-implant mucosa replication-A clinical study. Clin Oral Implants Res. 2022 Jun;33(6):598-606. doi: 10.1111/clr.13921. Epub 2022 Mar 26. PMID 35290685
- [Background] Monaco C, Scheda L, Baldissara P, Zucchelli G. Implant Digital Impression in the Esthetic Area. J Prosthodont. 2019 Jun;28(5):536-540. doi: 10.1111/jopr.12991. Epub 2018 Dec 3. PMID 30357992